CLINICAL TRIAL: NCT01351961
Title: Arterial Function and Structure and Evolution of Cognitive Impairment in Elderly Hypertensive Subjects With Subjective Memory Complaints
Brief Title: Vascular Alteration and Evolution of Cognitive Impairment
Acronym: ADELAHYDE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Athanase BENETOS, Coordinating Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-A01399-30
Record Dates: First submitted 2011-04-22; First posted 2011-05-11 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Impairment
Keywords: Hypertension; Cognitive function
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension | interventions — Blood Specimen Collection; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elderly hypertensive patients with mnemonic subjective (Other): Elderly hypertensive patients with mnemonic subjective without dementia. Interventions :
  blood sampling brain MRI Assessment of cognitive functions brain MRI and TEP cerebral Electrocardiogram and blood pressure Pulse wave velocity Quality of life questionnaire Urine sample Vascular explorations
  Interventions: Biological: blood sampling; Procedure: brain MRI and TEP cerebral; Other: Assessment of cognitive functions; Other: Electrocardiogram and blood pressure; Procedure: Vascular explorations; Biological: Urine sample

INTERVENTIONS:
Biological: blood sampling — take a sample of blood, 46 ml
Procedure: brain MRI and TEP cerebral — magnetic resonance imaging
Other: Assessment of cognitive functions — Folstein MMSE, Mac Nair scale, Depression (GDS) scale, The Benton Visual Retention Test, Test of verbal fluency, formal and categorical, Trail Making Test, Grober et Buschke scale (RL/RI-16), Apathy Robert scale, Praxis rating Scale .
Other: Electrocardiogram and blood pressure — Electrocardiogramm Blood pressure monitoring
Procedure: Vascular explorations — Pulse wave velocity, VWF, IMT
Biological: Urine sample

SUMMARY:
In the cross sectional study "Adelahyde 1" which took place between 2001 and 2005, the investigators data suggest that vascular alterations may play a role in the setting of subjective memory complaints.

This longitudinal study (Adelahyde 2) aims to confirm the role of vascular factors in the evolution of cognitive function and dementia.

DETAILED DESCRIPTION:
Background: The role of arterial hypertension and vascular alterations in the development of cognitive decline is a major issue in both research and clinical practice. In a recently published cross-sectional study (Kearney-Schwartz, Rossignol et al. 2009), conducted on the "ADELAHYDE" cohort comprised of older hypertensive patients with memory complaints, the investigators showed the association of arterial changes (hypertrophy and arterial stiffness, endothelial dysfunction) with cognitive functions and/or white matter hyperintensities on MRI. A longitudinal study is the only means to confirm the role of vascular factors in the evolution of cognitive function and onset of dementia.

Objectives: i) Primary: To establish, in the "ADELAHYDE" cohort, the relationship between vascular alterations assessed at baseline during the cross-sectional study (hypertrophy and arterial stiffness, endothelial dysfunction) and the evolution of cognitive function (primary study endpoint) over a 8-year follow-up period; ii) Secondary a) To investigate the evolution of white matter hyperintensities on MRI (secondary study endpoint) as a function of peripheral vascular status, and especially of endothelial function. b) Determine the role of genetic factors and biomarkers of oxidative stress (from DNA and serum biobanks collected at the first visit) in the evolution of cognitive functions and white matter hyperintensities.

Methods: Prospective longitudinal single center study. All patients (378 subjects) who participated in the baseline cross-sectional study conducted between 2001 and 2005, will be reconvened at the Clinical Investigation Centre (CIC) of Nancy.

As in the cross-sectional study, the following will be assessed in this longitudinal phase: pulse wave velocity (PWV), carotid ultrasonography, flow-mediated dilation, brain MRI with semi-quantification of white matter hyperintensities, cognitive function evaluation and measurement of various biomarkers of endothelial function.

Expected fallouts: A major benefit of this project is that this cohort has already been explored in terms of cognitive function, arterial properties and neurovascular imaging (MRI). Thus, the programmed reconvening of these subjects for this project in 2011 will enable us to identify the role of vascular alterations in the evolution of cognitive function and leucoaraiosis in this population at high risk of dementia over a period of at least 8 years. Finally, it could pave the way for further investigations, notably in the field of cognitive impairment prevention, aimed at reducing or delaying the onset of dementia by acting on the "vascular factor", which is potentially modifiable.

ELIGIBILITY:
Inclusion Criteria:

* patient who have participated Adelahyde 1 study
* patient who have signed a consent
* patient who have a social security

Exclusion Criteria:

* patient who can't understand information letter and who is not under legal protection

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Global memory, visual retention and verbal fluency composite score | up to two years

SECONDARY OUTCOMES:
vascular exploration | up to two years
  Pulse wave velocity, VWF, IMT
white matter hyperintensities by fazekas score. | up to two years
  Hyperintensities of white matter will be classified following the Fazekas scale (6 ranks.

CONTACTS AND LOCATIONS:
Overall Officials: Athanase BENETOS, professor, Principal Investigator — CHU NANCY
Locations (1):
- Chu Nancy, Nancy, France

REFERENCES:
- [Background] Ferreira JP, Kearney Schwartz A, Watfa G, Zohra L, Felblinger J, Boivin JM, Bracard S, Hossu G, Verger A, Joly L, Zannad F, Rossignol P, Benetos A. Memory Alterations and White Matter Hyperintensities in Elderly Patients With Hypertension: The ADELAHYDE-2 Study. J Am Med Dir Assoc. 2017 May 1;18(5):451.e13-451.e25. doi: 10.1016/j.jamda.2017.01.008. Epub 2017 Mar 6. PMID 28279605